CLINICAL TRIAL: NCT03192566
Title: The Pharmacokinetics of Intravenous Acetaminophen and Its Metabolites in Obese Children and Adolescents
Brief Title: Acetaminophen Dosing in Obese Adolescents
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: financial
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Janelle Vaughns, Principal Investigator, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00004651
Record Dates: First submitted 2017-05-28; First posted 2017-06-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Childhood
Keywords: Acetaminophen; Anesthesia; Adolescent; Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Determine the single dose pharmacokinetics of acetaminophen and its metabolites (glucuronide, sulphate, cystein and mercapturic acid) in obese children and adolescents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tylenol Dosing (Experimental): Dosing of Tylenol for postoperative pain relief will include:
  children < 16 years; 650 mg every 6 hours, max 2.6 gram per 24 hours and children > or equal to 16 years every 6 hours 1 g of acetaminophen, max 4 gram per 24 hours).
  Interventions: Drug: Tylenol

INTERVENTIONS:
Drug: Tylenol — Dosing of Tylenol for post operative pain control

SUMMARY:
Although there are numerous studies investigating the pharmacokinetic properties of intravenous acetaminophen in infants and children with normal weight, there are none in the obese pediatric patient . This study will investigate the pharmacokinetics and pharmacodynamics of acetaminophen (total Cl and Vd) in obese children and adolescents

DETAILED DESCRIPTION:
Obesity represents one of the most important public health issues according to the World Health Organization. It has reached epidemic proportions globally, with approximately 1.5 billion overweight adults aged 20 years and older and at least 600 million of them clinically obese .Childhood obesity is particularly problematic, because the co morbid disease states which accompany early obesity may require frequent pharmacotherapy and/or surgical intervention. Many of the metabolic and cardiovascular complications of obesity may also be present during childhood. Despite increased pharmacotherapy among obese patients, there is a paucity of dosing guidelines for this population. Optimal drug dosing in obese pediatric patients has not been explored as the present data available is specific for obese adults. Acetaminophen is one of the most commonly used medications in pediatric patients.

Although there are numerous studies investigating the pharmacokinetic properties of intravenous acetaminophen in infants and children with normal weight there are none in the obese pediatric patient . This study will investigate the pharmacokinetics and pharmacodynamics of acetaminophen (total clearance and volume of distribution in obese children and adolescents

ELIGIBILITY:
Inclusion Criteria:

* Participant will be a Children's National Health System (CNHS) inpatient or outpatient admitted for at least 24 hours observation as part of the surgical plan of care.
* Age range will be between 10 and 18.
* BMI% will be calculated using height and weight and will include the 5th-85th% (normal weight) and greater than or equal to 95th %.( obese weight)
* ASA physical classification of I, II or III.
* All racial and ethnic groups will be included

Exclusion Criteria:

* Any patient that is pregnant or lactating.
* Renal insufficiency identified by GFR <60 ml/min/1.73m2 and/or creatinine > 3 times upper limit of normal values
* Liver disease identified by : AST, ALT, γ-GT, bilirubin, albumin and AlkP and PT > 3 times upper limit of normal values
* Patients with Gilbert-Meulengracht Syndrome
* Chronic alcohol intake or use of alcohol within last 72 hours
* Patients who are treated with drugs know to effect CYP2E1(inhibition: dithiocarb and disulfiram. Induction: isoniazid) and UGT (UDP-glucuronyltransferases) (induction: estradiol-containing contraceptives, carbamazepine, phenobarbital, phenytoin, mesuximide, oxcarbazepine, rifampicin, primidone, atazanavir / ritonavir, lopinavir / ritonavir, olanzapine, retigabine , nevaripine, efavirenz, saquinavir, nelfinavir, lamotrigine, felbamate, zonisamide, bupropion. Inhibition: valproic acid)
* Diabetes mellitus type II patients
* Smoking
* Acetaminophen intake up to 24 hours before enrollment.
* Acetaminophen allergy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Systemic clearance of acetaminophen and its metabolites (glucuronide, sulphate, cystein and mercapturic acid) in adolescent surgical patients | up to 3 years

SECONDARY OUTCOMES:
Evaluate postoperative pain management using the numerical rating scale system. | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Result] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Result] Cali AM, Caprio S. Obesity in children and adolescents. J Clin Endocrinol Metab. 2008 Nov;93(11 Suppl 1):S31-6. doi: 10.1210/jc.2008-1363. PMID 18987268
- [Result] Erstad BL. Which weight for weight-based dosage regimens in obese patients? Am J Health Syst Pharm. 2002 Nov 1;59(21):2105-10. doi: 10.1093/ajhp/59.21.2105. No abstract available. PMID 12434728
- [Result] Blouin RA, Warren GW. Pharmacokinetic considerations in obesity. J Pharm Sci. 1999 Jan;88(1):1-7. doi: 10.1021/js980173a. No abstract available. PMID 9874695
- [Result] Cheymol G. Clinical pharmacokinetics of drugs in obesity. An update. Clin Pharmacokinet. 1993 Aug;25(2):103-14. doi: 10.2165/00003088-199325020-00003. PMID 8403734
- [Result] Mohammed BS, Engelhardt T, Cameron GA, Cameron L, Hawksworth GM, Hawwa AF, McElnay J, Helms PJ, McLay JS. Population pharmacokinetics of single-dose intravenous paracetamol in children. Br J Anaesth. 2012 May;108(5):823-9. doi: 10.1093/bja/aes025. Epub 2012 Mar 1. PMID 22389380
- [Result] Zuppa AF, Hammer GB, Barrett JS, Kenney BF, Kassir N, Mouksassi S, Royal MA. Safety and population pharmacokinetic analysis of intravenous acetaminophen in neonates, infants, children, and adolescents with pain or Fever. J Pediatr Pharmacol Ther. 2011 Oct;16(4):246-61. doi: 10.5863/1551-6776-16.4.246. PMID 22768009